CLINICAL TRIAL: NCT00031668
Title: A Phase III Study of Involved Field Radiation Therapy (IFRT) in Patients With Histologically Aggressive Non-Hodgkin's Lymphoma Following High Dose Chemotherapy and Autologous Hematopoietic Stem Cell Transplantation (ASCT)
Brief Title: Radiation Therapy in Relapsed or Refractory Non-Hodgkin's Lymphoma Who Have Undergone Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: LY8; CAN-NCIC-LY8; CDR0000069214 (Other: PDQ)
Record Dates: First submitted 2002-03-08; First posted 2003-07-01 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia; recurrent adult diffuse large cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult T-cell leukemia/lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known if giving radiation therapy after stem cell transplantation is more effective than stem cell transplantation alone in treating relapsed or refractory non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to determine the effectiveness of radiation therapy in treating patients who have relapsed or refractory non-Hodgkin's lymphoma and have undergone autologous stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the 3-year progression-free survival of patients with relapsed or refractory aggressive non-Hodgkin's lymphoma treated with high-dose chemotherapy and autologous hematopoietic stem cell transplantation with or without involved-field radiotherapy.
* Compare the overall survival of patients treated with these regimens.
* Compare 3-year progression-free disease within and outside radiotherapy fields in patients treated with these regimens.
* Compare quality of life of patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to response to pre-salvage chemotherapy (primary refractory disease vs relapse), response to post-salvage chemotherapy (complete/unconfirmed complete vs partial), and participating center. Within 6-8 weeks after completion of autologous hematopoietic stem cell transplantation, patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo involved-field radiotherapy (IFRT) 5 days a week for 3-5 weeks in the absence of unacceptable toxicity.
* Arm II: Patients undergo observation only. Quality of life in arm I is assessed at baseline, on day 1 of IFRT, at weeks 2 and 4 during IFRT, at 1 month, 4 months, every 3 months for 2 years, every 6 months for 1 year, and then annually for 2 years. Quality of life in arm II is assessed at baseline, 1 month, 2 months, every 3 months for 2 years, every 6 months for 1 year, and then annually for 2 years.

Patients are followed at 1 month, every 3 months for 2 years, every 6 months for 1 year, and then annually for 2 years.

PROJECTED ACCRUAL: A total of 230 patients (115 per treatment arm) will be accrued for this study within 4.2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma

  * Diffuse large cell lymphoma, B-cell (includes primary mediastinal B-cell lymphoma and T-cell rich B-cell lymphoma)
  * Previous indolent lymphoma (follicular center cell lymphoma, marginal zone lymphoma, including extranodal MALT lymphoma and lymphoplasmacytoid lymphoma) with transformation to diffuse large B-cell lymphoma at relapse
  * Peripheral T-cell lymphoma
  * Anaplastic large cell lymphoma (T cell or null cell)
  * Small non-cleaved Burkitt-like lymphoma
* Relapsed or refractory disease after first-line anthracycline-based chemotherapy

  * Bulky disease, nodal or extranodal

    * Clinically or radiographically measurable mass at least 5 cm in diameter OR
  * Non-bulky disease, nodal or extranodal, excluding diffuse organ (lung, liver, kidney, or bone marrow) involvement

    * Clinically or radiographically measurable disease more than 1.5 cm in greatest transverse diameter
* Biopsy at relapse not required except for transformed lymphomas

  * Patients with transformed lymphoma at diagnosis, but with indolent histology without transformation at relapse, are not eligible
* No patients with stage IA or IIA disease at initial diagnosis who, at time of relapse or diagnosis of refractory disease prior to salvage therapy, remained in stage IA or IIA, with no new disease sites, without having received radiotherapy
* Received up to 2 regimens and 4 courses of salvage chemotherapy

  * Monoclonal antibodies (e.g., rituximab) are not considered salvage chemotherapy
  * Achieved complete response (CR), unconfirmed CR, or partial response (PR) if bulky disease OR
  * Achieved PR (but not CR) if non-bulky disease
* No residual disease involving extranodal organs diffusely (e.g., liver, lung, bone, kidney, or leptomeningeal) after salvage chemotherapy
* Planned autologous hematopoietic stem cell transplantation (ASCT)

  * ASCT conditioning must be with high-dose BEAM (carmustine, etoposide, cytarabine, and melphalan) chemotherapy
* No disease progression after ASCT
* No major organ complication or poor hematologic recovery from ASCT that would preclude initiation of study radiotherapy within 14 weeks after ASCT
* No more than 2 non-contiguous nodal or extranodal areas of bulky/residual disease requiring more than 2 separate involved-field radiotherapy volume arrangements (e.g., field arrangement covering up to 2 involved lymph node regions or extranodal sites, with or without 1 adjacent nodal/region or extranodal site)
* No active CNS lymphoma (parenchymal brain and/or leptomeningeal)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except basal cell carcinoma of the skin

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* No prior radioimmunotherapy

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior total body irradiation
* No prior radiotherapy to the site of bulky disease or residual tumor

Surgery:

* Not specified

Other:

* No other concurrent anti-cancer therapy unless documentation of disease progression

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2001-01-31 (Actual); Primary Completion 2009-02-10 (Actual); Study Completion 2009-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Tsang, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada
Locations (9):
- Canada (9):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No